CLINICAL TRIAL: NCT01720628
Title: The Relationship Between Serum Levels of Angiogenin, bFGF, VEGF and Ocular Involvement in Patients With Behçet's Disease
Status: Completed | Type: Observational
Sponsor: Turkish Ophthalmology Society (Other)
Responsible Party: Principal Investigator, Yeşim Gedik Oğuz, MD, Turkish Ophthalmology Society
Other Study IDs: AFV-5813
Record Dates: First submitted 2012-10-23; First posted 2012-11-02 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Behçet's Disease
Keywords: Angiogenin, Behçet's disease, bFGF, VEGF
MeSH Terms: conditions — Behcet Syndrome | interventions — Vascular Endothelial Growth Factor A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Behçet's patients: Serum levels of angiogenin, bFGF, VEGF levels in Behçet's patients with ocular involvement group, without ocular involvement group and control group
  Interventions: Other: serum levels of angiogenin, bFGF, VEGF

INTERVENTIONS:
Other: serum levels of angiogenin, bFGF, VEGF — Behçet's patients

SUMMARY:
Objectives: Behçet's disease (BD) is a systemic vasculitis. Since vascular endothelial dysfunction plays a prominent role in the pathogenesis of the disease, we considered angiogenic cytokines as an interesting target for investigation in BD. The aim of this study was to investigate the possible role of angiogenin, vascular endothelial growth factor (VEGF) and basic fibroblast growth factor (bFGF) in the pathogenesis of BD.

Design and Methods: Sixty five patients with BD and 21 healthy control subjects were included in the study. Serum angiogenin, bFGF and VEGF concentrations were determined by using in vitro enzyme immunoassay (ELISA) kits according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65
* fulfilling the international diagnostic criteria for Behçet's disease

Exclusion Criteria:

* to have another systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Turkish patients fulfilling the international diagnostic criteria for Behçet's disease
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Serum levels of angiogenin in Behçet's patients with or without ocular involvement | 1 year
  The median serum angiogenin level was significantly higher in all patients with BD than controls (P=0.001). However there was no statistically significant difference between all patients and patients with or without ocular involvement. The mean serum bFGF and the median serum VEGF levels were higher in patients with ocular involvement than all patients, patients without ocular involvement and controls. But these differences did not reach statistical significance.

SECONDARY OUTCOMES:
Serum levels of bFGF in Behçet's patients with or without ocular involvement | 1 year

OTHER OUTCOMES:
Serum levels of VEGF in Behçet's patients with or without ocular involvement | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: ali yalçındağ, Study Director — * Dışkapı Yıldırım Beyazıt Training and Research Hospital, Department of Clinical Biochemistry
Locations (1):
- Ankara University, Faculty of Medicine, Department of Ophthalmology, Ankara, Turkey (Türkiye)